CLINICAL TRIAL: NCT05559268
Title: Single Dose Subcutaneous Injections of Denosumab for Patients Underwent Cemented Total Knee Arthroplasty. A Randomized Controlled Study on the Effects on Bone Microarchitecture, Skeletal Muscle, Cartilage and Synovium
Brief Title: Effects of Denosumab on Bone Microarchitecture After Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Xiang Shuai, MD, Dr., The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Denosumab AHQD
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental)
  Interventions: Drug: Denosumab 60 MG/ML Injectable Solution [Prolia]
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab 60 MG/ML Injectable Solution [Prolia] — 1 ml (60 mg) subcutaneous injection Denosumab give in the posterior part of the upper arm after TKA
  Arms: Denosumab
Drug: Placebo — 1 ml (60 mg) subcutaneous injection Saline give in the posterior part of the upper arm after TKA
  Arms: Placebo

SUMMARY:
This study evaluates single dose of Denosumab in decreasing systemic and periprosthetic bone resorption after Total Knee Arthroplasty compared to placebo in 60 patients (30 placebo and 30 Denosumab) within 2 months after surgery. This study also evaluates the anti-RANKL effect of single dose of Denosumab in serum, skeletal muscle, synovium, fat, and cartilage.

ELIGIBILITY:
Inclusion Criteria:

Patients with Bilateral Knee Osteoarthritis treated with Staged Bilateral Total Knee Arthroplasty, with an Interval of 8 weeks

Exclusion Criteria:

Patients allergies to Denosumab Patients with previous Osteoporosis treatment Patients with renal failure Patients with previous Bisphosphonate treatment for more than 5 years Patients failed to finish contralateral Total Knee Arthroplasty at 8 weeks

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Bone Microarchitecture | 8 weeks
  Bone Microarchitecture on microCT
Bone turnover markers | 8 weeks
  βCTXI, NTXI, 25(OH)VD3, CT, BGP, PINP

SECONDARY OUTCOMES:
intermuscular and intramuscular adipose | 8 weeks
  intermuscular and intramuscular adipose on biopsy slice
Mankin Histological-Histochemical Grading of Cartilage | 8 weeks
  Mankin Histological-Histochemical Grading of Cartilage
Histopathological grading of synovium | 8 weeks
  Histopathological grading of synovium

OTHER OUTCOMES:
Certain protein expression in bone, muscle, synovium and cartilage | 8 weeks
  Certain protein expression in bone, muscle, synovium and cartilage

IPD SHARING:
Plan to Share IPD: Undecided